CLINICAL TRIAL: NCT04814771
Title: Mass Balance Recovery, Pharmacokinetics, Metabolite Identification and Profiling of 14C-labeled TS-142 in Healthy Adult Subjects.
Brief Title: Mass Balance Study of TS-142 in Healthy Adult Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TS142-206
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2021-06

CONDITIONS: Healthy Male Subjects
MeSH Terms: interventions — TS-142

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [14C] TS-142 (Experimental): Participants will receive oral [14C] TS-142 under fasted conditions
  Interventions: Drug: [14C] TS-142

INTERVENTIONS:
Drug: [14C] TS-142 — Subjects received single dose of 7.5 mg of TS-142 containing 20 kBq [14C]TS-142 as an oral solution

SUMMARY:
To assess the plasma pharmacokinetics, the routes extent of elimination, and the metabolites of TS-142 after single oral dose of [14C] TS-142 in Japanese healthy male subjects.

To assess the safety of single oral dose of [14C] TS-142 in Japanese healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Japanese males aged >=20 and <40 years at the signing of informed consent
* Subjects whose body mass index (BMI) >=18.5 and <25.0 kg/m2 at screening
* Subjects who have no abnormal findings in the physical examination, vital signs, and standard 12-lead ECG in the screening test and the test on the day of admission and the test obtained prior to administration of the investigational drug, and whose clinical test results are within the standard values of the clinical trial site in the screening test and the test on the day of admission. However, if who showed abnormal findings but not clinically significant, they can be enrolled in clinical trials based on comprehensive consideration of medical viewpoints by the principal investigator(s) or subinvestigator(s).
* Subjects who understand, and have willingness and ability to read and sign, the informed consent form

Exclusion Criteria:

* Subjects who have received a substance labeled with a radioisotope within the last 12 months prior to dosing of the investigational drug
* Subjects who have been exposed to a large amount of radiation for therapeutic or diagnostic reasons (CT scan, stomach X-ray, PET scan etc.) within the last 12 months prior to dosing of the investigational drug
* Occupationally exposed worker in the last 12 months prior to dosing of the investigational drug
* Subjects who have had 3 days or less that one or more spontaneous defecations (defecation that occurs without laxatives, enemas, disimpaction) within 7 days before consent is obtained and during the 7 days until on the day of admission. Those who have diarrhea during the 7 days until on the day of admission
* History of any disease or surgery which have impact on investigational drug absorption such as gastrectomy, gastroenterostomy or bowel resection
* Other protocol defined exclusion criteria could apply

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Radioactivity concentration in whole blood and plasma | Up to 168 hours after dosing
Calculation of cumulative urinary and fecal recovery of total radioactivity, and calculation of mass balance as a sum of the percentages of total radioactivity recovered in urine and faeces | Up to 168 hours after dosing
Concentration of unchanged form and its major metabolites in plasma | Up to 168 hours after dosing
Percentage of TS-142 and metabolites to total radioactivity in plasma | Up to 168 hours after dosing
Percentage of TS-142 and metabolites to total radioactivity in urine and faeces | Up to 168 hours after dosing
Metabolite profiling and structural identification of metabolites in plasma, urine and faeces | Up to 168 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Direcoter, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- Taisho Pharmaceutical Co., Ltd selected site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No